CLINICAL TRIAL: NCT04860570
Title: Retrospective, Multi-centric Study Comparing the Incidence of Surgical Site Infections in Patients Receiving Open Appendectomy With Double-ring Wound-edge Protectors Versus Laparoscopic Appendectomy
Brief Title: Are Double-ring Wound-edge Protectors Effective for Preventing Superficial Surgical Site Infection After Open Appendectomy?
Acronym: sSSI-2RWEPs
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital Medina del Campo (Other)
Responsible Party: Principal Investigator, Johnn Henry Herrera Kok, Dr. Johnn Henry Herrera Kok, Hospital Medina del Campo
Other Study IDs: PI 21-2140 MEDINA
Record Dates: First submitted 2021-04-22; First posted 2021-04-27 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-12

CONDITIONS: Acute Appendicitis; Surgical Site Infection
Keywords: Acute appendicitis; double-ring wound-edge protector; superficial surgical site infection
MeSH Terms: conditions — Appendicitis; Surgical Wound Infection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Open Appendectomy (OA) + Double-ring wound-edge protector (2RWEP): Intervention group: Patients with diagnosis of acute appendicitis treated by open appendectomy using a double-ring wound-edge protector.
  Interventions: Device: Double-ring wound-edge protector
- Laparoscopic Appendectomy (LA): Control group: Patients with diagnosis of acute appendicitis treated by laparoscopic appendectomy.

INTERVENTIONS:
Device: Double-ring wound-edge protector — Double-ring wound-edge protector: Alexis Applied Medical ®, Rancho Santa Margarita, California.
  Groups: Open Appendectomy (OA) + Double-ring wound-edge protector (2RWEP)

SUMMARY:
This study aims to evaluate the utility of double-ring wound-edge protectors to prevent the development of superficial surgical site infections after open appendectomy.

DETAILED DESCRIPTION:
This is a multi-centric retrospective study comparing patients of similar characteristics with diagnosis of acute appendicitis that have been treated either by open appendectomy using a double-ring wound-edge protector or by laparoscopic appendectomy between January 2011 and December 2016 at Hospital Recoletas Campo Grande de Valladolid and Hospital Comarcal de Medina del Campo.

The main objective of the study is to compare the incidence of superficial surgical site infection in both groups.

All patients included in the study must meet inclusion criteria and all data will be collected anonymously in order to comply with local law on personal data protection (Organic Law 15/1999 from 13 December about personal data protection).

The authors of the study expect results of the study to be comparable with those in current literature regarding surgical site infections, hospital stay and procedure safety.

ELIGIBILITY:
Inclusion Criteria:

* Age of at least 15 years old.
* Clinical diagnosis of acute appendicitis.
* Treated by: Open appendectomy + double-ring wound-edge protector or Laparoscopic appendectomy.
* Note: with the aim of avoiding selection bias, all patients presenting risk factors for surgical site infections (eg obesity, diabetes, malnourishment, immunosupression, etc.) will be included in the present study.

Exclusion Criteria:

* Patients who did not receive prophylactic antibiotic.
* Source of abdominal pathology other than the caecal appendix.
* Follow-up period less than 30 days.

Ages: 15 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All patients 15 years old or older, with diagnosis of acute appendicitis who were treated either by open appendectomy using a double-ring wound-edge protector or by laparoscopic appendectomy at Hospital Recoletas Campo Grande de Valladolid and Hospital Comarcal de Medina del Campo.
Sampling Method: Probability Sample
Enrollment: 671 (Estimated)
Dates: Start 2024-10-25 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Superficial surgical site infection (sSSI) | 30 days after surgery
  To compare the incidence of sSSI in both groups (OA+2RWEP versus LA) during postoperative period to determine wether 2RWEP are useful in reducing sSSI after open appendectomy.

SECONDARY OUTCOMES:
Organ-space surgical site infection (oeSSI) | 30 days
  To compare the incidence of oeSSI in both groups (OA+2RWEP versus LA) during postoperative period to determine wether 2RWEP are useful in reducing oeSSI after open appendectomy.
Hospital stay | 30 days
  To compare the length of hospital stay in both groups (OA+2RWEP versus LA) to determine wether 2RWEP are useful in reducing hospital stay.

CONTACTS AND LOCATIONS:
Overall Officials: Johnn Henry Herrera Kok, Principal Investigator — Complejo Asistencial Universitario de León, Spain
Locations (1):
- Hospital Comarcal de Medina del Campo, Medina del Campo, Spain

IPD SHARING:
Plan to Share IPD: No